

| Official Title: | Randomized Trial of Trust in Online Videos About Prostate Cancer |
|---|---|
| NCT Number: | NCT05886751 |
| Study Number: | 20-00540 |
| Document Type: | Informed Consent Form |
| Date of the Document: | • May 29, 2021 |

Study: #S20-00540 Version: 05/21/2021

## ELECTRONIC CONSENT FOR ONLINE SURVEY

Thank you for your interest in this study about online health videos!

We are asking you to participate in this study because you are an adult living in the United States who uses the internet. The purpose of this project is to understand the perspective of U.S. adults on different videos about prostate cancer. Results from this study will be used to inform the creation of future videos about health.

If you agree to participate in this study, you will be asked to follow the embedded link to an anonymous survey that will take approximately 15 minutes to complete. The survey will include questions about demographics and internet use. It will also include an embedded video about prostate cancer and ask a series of questions about your reaction to the video. The survey will not ask for your name or any other personally identifiable information; your answers will be anonymous. Once you've watched the video and completed the survey, your participation in the study is complete.

This study is funded by the Department of Defense (DoD). The confidentiality section allows the DoD access to research records as a part of its human subjects protection oversight activities. The risks of participating in this study are minimal. While there are no physical risks involved, there is a small risk of a breach of confidentiality, however, multiple safeguards are in place to ensure information security. There will be no direct benefit to you from participating in this study. We hope that the results will help the public in the future by informing the creation of educational materials about prostate cancer.

Your participation in this study is completely voluntary; you do not have to participate in this study unless you want to. Your decision whether or not to participate in this study will not affect your medical care. If you decide to take part in this study, you must provide an answer for each question in the survey, however you are free to withdraw from the study at any time by exiting the survey. Once you complete the survey, you will receive your standard incentive from Dynata. There will be no cost to you for being in this study.

If a member of the research team cannot be reached or you want to talk to someone other than those working

For more information or questions about this study, please contact the study coordinators:

on the study, you may contact the Institutional Review Board (IRB) at (212) 263-4110.

| Many | thanks in advance for your participation! |
|---|---|
| | I have read the above and understand that my participation is voluntary and I |
| | AGREE TO PARTICIPATE in this study. I have read the above and DO NOT WISH to take part in this study |